CLINICAL TRIAL: NCT03592745
Title: Evaluating the Use of Transcutaneous Vagus Nerve Stimulation (tVNS) and Robotic Training to Improve Upper Limb Motor Recovery After Stroke
Brief Title: Transcutaneous Vagus Nerve Stimulation (tVNS) and Robotic Training to Improve Arm Function After Stroke
Acronym: tVNS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Bruce Volpe, Principal Investigator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-0404
Record Dates: First submitted 2018-07-05; First posted 2018-07-19 (Actual); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-05

CONDITIONS: Stroke; Cerebrovascular Accident (CVA); Hemiparesis
Keywords: Transcutaneous vagus nerve stimulation (tVNS); VNS; robotic therapy; occupational therapy; motor rehabilitation
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: This is a double-blind, sham controlled treatment study in which patients will have a 50/50 chance of receiving robotic arm therapy with either active transcutaneous vagus nerve stimulation (tVNS) or sham tVNS (placebo).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both the participants and investigators performing and analyzing clinical and objective outcome measures will remain blind to condition. Participants will be told that they have a 50-50 chance of receiving either active or sham stimulation, but they will not be told which condition they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- active tVNS + robotic arm therapy (Experimental): Transcutaneous Vagus Nerve Stimulation (tVNS) will be delivered non-invasively via the ear (targeting the auricular branch of the vagus nerve) during robotic arm therapy sessions lasting ~60 minutes, 3x per week for 3 weeks.
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation (tVNS)
- sham tVNS + robotic arm therapy (Sham Comparator): Sham (placebo) transcutaneous Vagus Nerve Stimulation (tVNS) will be delivered non-invasively via the ear (targeting the auricular branch of the vagus nerve) during robotic arm therapy sessions lasting ~60 minutes, 3x per week for 3 weeks.
  Interventions: Device: Sham Transcutaneous Vagus Nerve Stimulation (tVNS)

INTERVENTIONS:
Device: Transcutaneous Vagus Nerve Stimulation (tVNS) — tVNS is a non-invasive form of vagus nerve stimulation, activating the auricular branch of the vagus nerve transcutaneously through the cymba concha at the pinna of the ear.
  Other Names: Transauricular Vagus Nerve Stimulation
  Arms: active tVNS + robotic arm therapy
Device: Sham Transcutaneous Vagus Nerve Stimulation (tVNS) — tVNS is a non-invasive form of vagus nerve stimulation, activating the auricular branch of the vagus nerve transcutaneously through the cymba concha at the pinna of the ear. Sham tVNS means the patient is wearing the device, but it is turned off and not delivering current during the treatment. This is a placebo condition, which is used as a study control.
  Other Names: Sham Transauricular Vagus Nerve Stimulation
  Arms: sham tVNS + robotic arm therapy

SUMMARY:
The purpose of this study is to evaluate if multiple therapy sessions of Transcutaneous Vagus Nerve Stimulation (tVNS) combined with robotic arm therapy lead to a greater functional recovery in upper limb mobility after stroke than that provided by robotic arm therapy in a sham stimulation condition.

DETAILED DESCRIPTION:
Promising new animal research suggests that vagus nerve stimulation paired with motor intervention induces movement-specific plasticity in the motor cortex and improves limb function after stroke. These results were recently extended to the first clinical trial, in which patients with stroke demonstrated significant improvements in upper limb function following rehabilitation paired with implanted VNS. Currently, vagus nerve stimulation is being used clinically to treat a number of human diseases including migraine headaches, epilepsy, and depression, and these investigations are expanding to deliver stimulation via a transcutaneous route to potentially improve intervention efficacy and decrease side effects. This pilot study will combine non-invasive transcutaneous stimulation of the vagus nerve with upper limb robotic therapy to investigate the potential of tVNS to augment improvements gained with robotic therapy in patients with chronic hemiparesis after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18 and 85 years of age
* First single focal unilateral supratentorial ischemic stroke with diagnosis verified by brain imaging (MRI or CT scans) that occurred at least 6 months prior
* Cognitive function sufficient to understand the experiments and follow instructions (per interview with Speech Pathologist or PI)
* Fugl-Meyer assessment 12 to 44 out of 66 (neither hemiplegic nor fully recovered motor function in the muscles of the shoulder, elbow, and wrist).

Exclusion Criteria:

* Botox treatment within 3 months of enrollment
* Fixed contraction deformity in the affected limb
* Complete and total flaccid paralysis of all shoulder and elbow motor performance
* Prior injury to the vagus nerve
* Severe dysphagia
* Introduction of any new rehabilitation interventions during study
* Individuals with scar tissue, broken skin, or irremovable metal piercings that may interfere with the stimulation or the stimulation device
* Highly conductive metal in any part of the body, including metal injury to the eye; this will be reviewed on a case by case basis for PI to make a determination
* Pregnant or plan on becoming pregnant or breastfeeding during the study period
* Significant arrhythmias, including but not limited to, atrial fibrillation, atrial flutter, sick sinus syndrome, and A-V blocks (enrollment to be determined by PI review)
* Presence of an electrically, magnetically or mechanically activated implant (including cardiac pacemaker), an intracerebral vascular clip, or any other electrically sensitive support system; Loop recorders will be reviewed on a case by case basis by PI and the treating Cardiologist to make a determination

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Feinstein Institute for Medical Research, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dawson J, Pierce D, Dixit A, Kimberley TJ, Robertson M, Tarver B, Hilmi O, McLean J, Forbes K, Kilgard MP, Rennaker RL, Cramer SC, Walters M, Engineer N. Safety, Feasibility, and Efficacy of Vagus Nerve Stimulation Paired With Upper-Limb Rehabilitation After Ischemic Stroke. Stroke. 2016 Jan;47(1):143-50. doi: 10.1161/STROKEAHA.115.010477. Epub 2015 Dec 8. PMID 26645257
- [Background] Capone F, Miccinilli S, Pellegrino G, Zollo L, Simonetti D, Bressi F, Florio L, Ranieri F, Falato E, Di Santo A, Pepe A, Guglielmelli E, Sterzi S, Di Lazzaro V. Transcutaneous Vagus Nerve Stimulation Combined with Robotic Rehabilitation Improves Upper Limb Function after Stroke. Neural Plast. 2017;2017:7876507. doi: 10.1155/2017/7876507. Epub 2017 Dec 10. PMID 29375915
- [Background] Khodaparast N, Hays SA, Sloan AM, Fayyaz T, Hulsey DR, Rennaker RL 2nd, Kilgard MP. Vagus nerve stimulation delivered during motor rehabilitation improves recovery in a rat model of stroke. Neurorehabil Neural Repair. 2014 Sep;28(7):698-706. doi: 10.1177/1545968314521006. Epub 2014 Feb 18. PMID 24553102
- [Background] Khodaparast N, Hays SA, Sloan AM, Hulsey DR, Ruiz A, Pantoja M, Rennaker RL 2nd, Kilgard MP. Vagus nerve stimulation during rehabilitative training improves forelimb strength following ischemic stroke. Neurobiol Dis. 2013 Dec;60:80-8. doi: 10.1016/j.nbd.2013.08.002. Epub 2013 Aug 15. PMID 23954448
- [Background] Hays SA. Enhancing Rehabilitative Therapies with Vagus Nerve Stimulation. Neurotherapeutics. 2016 Apr;13(2):382-94. doi: 10.1007/s13311-015-0417-z. PMID 26671658
- [Background] Volpe BT, Huerta PT, Zipse JL, Rykman A, Edwards D, Dipietro L, Hogan N, Krebs HI. Robotic devices as therapeutic and diagnostic tools for stroke recovery. Arch Neurol. 2009 Sep;66(9):1086-90. doi: 10.1001/archneurol.2009.182. PMID 19752297
- [Derived] Chang JL, Coggins AN, Saul M, Paget-Blanc A, Straka M, Wright J, Datta-Chaudhuri T, Zanos S, Volpe BT. Transcutaneous Auricular Vagus Nerve Stimulation (tAVNS) Delivered During Upper Limb Interactive Robotic Training Demonstrates Novel Antagonist Control for Reaching Movements Following Stroke. Front Neurosci. 2021 Nov 25;15:767302. doi: 10.3389/fnins.2021.767302. eCollection 2021. PMID 34899170

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active tVNS + Robotic Arm Therapy | Sham tVNS + Robotic Arm Therapy
Started | 18 | 18
Completed | 15 | 15
Not Completed | 3 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — study temporary closure due to covid-19 pandemic | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tVNS + Robotic Arm Therapy | Sham tVNS + Robotic Arm Therapy | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Full Range); unit: years] | 56.0 [27.9 to 81.1] | 62.0 [45.9 to 75.6] | 59.0 [27.9 to 81.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 7 | 10 | 17
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Median Absolute Change From Baseline in Electromyographic (EMG) Peak Amplitude of the Bicep/Tricep
Description: The median absolute change in surface electromyographic (sEMG) peak amplitude of the bicep/tricep during gravity-eliminated, unassisted extensor movements was calculated from baseline to discharge at 3 weeks (immediately following the intervention) and again at 16 weeks (3 months follow-up from the intervention) in each training condition (sham tVNS + robotic arm training vs. active tVNS + robotic arm training). Bicep and tricep peak sEMG amplitude scores were calculated as a percentage of the maximal volitional contraction (MVC), with larger values indicating a greater absolute change (negative or positive) in bicep/tricep peak muscle activity during extensor movements.
Time Frame: baseline, discharge at 3 weeks (immediately following the intervention), and follow-up at 16 weeks (3 months after the intervention)
Population: 30 patients completed 9 sessions (3x/week for 3 weeks) of robotic arm training + sham or active tVNS, and 3 month follow-up at 16 weeks. One patient in the sham condition had corrupted sEMG measures, so 29 participants were consequently included in the efficacy analysis.
Measure: Median (Inter-Quartile Range); unit: percentage of MVC
Arm/Group | Active tVNS + Robotic Arm Therapy | Sham tVNS + Robotic Arm Therapy
Number analyzed (Participants) | 15 | 14
percentage of MVC
  Median absolute change in bicep peak amplitude from baseline to discharge after 3 weeks of training | 22.310 [16.780 to 32.630] | 7.010 [2.057 to 13.845]
  Median absolute change in tricep peak amplitude from baseline to discharge after 3 weeks of training | 16.070 [11.460 to 19.930] | 10.055 [5.330 to 32.553]
  Median absolute change in bicep peak amplitude from baseline to 3 month follow-up | 21.730 [3.240 to 33.850] | 13.545 [3.010 to 29.618]
  Median absolute change in tricep peak amplitude from baseline to 3 month follow-up | 10.520 [6.420 to 24.070] | 11.455 [7.303 to 18.848]
Statistical Analysis 1: Comparison: Active tVNS + Robotic Arm Therapy vs Sham tVNS + Robotic Arm Therapy; Test type: Equivalence — Statistical analysis of the median absolute change in bicep peak sEMG amplitude from baseline to DC immediately following 3 weeks of training was measured in the active vs. sham tVNS conditions. Null hypothesis is that there is no difference in median absolute change in bicep peak sEMG amplitude between the active and sham tVNS conditions. A significance level of 0.05 was used (two-tailed); p = 0.002, Wilcoxon (Mann-Whitney) — The Mann-Whitney Wilcoxon test was performed to compare median absolute change in bicep peak sEMG amplitude from baseline to 3 weeks (discharge) across two separate study conditions (active vs. sham tVNS); U value = 32.000
Statistical Analysis 2: Comparison: Active tVNS + Robotic Arm Therapy vs Sham tVNS + Robotic Arm Therapy; Test type: Equivalence — Statistical analysis of the median absolute change in tricep peak sEMG amplitude from baseline to DC immediately following 3 weeks of training was measured in the active vs. sham tVNS conditions. Null hypothesis is that there is no difference in median absolute change in bicep peak sEMG amplitude between the active and sham tVNS conditions. A significance level of 0.05 was used (two-tailed); p = 0.445, Wilcoxon (Mann-Whitney) — The Mann-Whitney Wilcoxon test was performed to compare median absolute change in tricep peak sEMG amplitude from baseline to 3 weeks (discharge) across two separate study conditions (active vs. sham tVNS); U value = 87.000
Statistical Analysis 3: Comparison: Active tVNS + Robotic Arm Therapy vs Sham tVNS + Robotic Arm Therapy; Test type: Equivalence — Statistical analysis of the median absolute change in bicep peak sEMG amplitude from baseline to week 16 (3 month follow-up after training) was measured in the active vs. sham tVNS conditions. Null hypothesis is that there is no difference in median absolute change in bicep peak sEMG amplitude between the active and sham tVNS conditions. A significance level of 0.05 was used (two-tailed); p = 0.678, Wilcoxon (Mann-Whitney) — The Mann-Whitney Wilcoxon test was performed to compare the median absolute change in bicep peak sEMG from baseline to 16 weeks (follow-up) across two separate study conditions (active vs. sham tVNS); U value = 95.000
Statistical Analysis 4: Comparison: Active tVNS + Robotic Arm Therapy vs Sham tVNS + Robotic Arm Therapy; Test type: Equivalence — Statistical analysis of the median absolute change in tricep peak sEMG amplitude from baseline to week 16 (3 month follow-up after training) was measured in the active vs. sham tVNS conditions. Null hypothesis is that there is no difference in median absolute change in bicep peak sEMG amplitude between the active and sham tVNS conditions. A significance level of 0.05 was used (two-tailed); p = 0.777, Wilcoxon (Mann-Whitney) — The Mann-Whitney Wilcoxon test was performed to compare the median absolute change in tricep peak sEMG from baseline to 16 weeks (follow-up) across two separate study conditions (active vs. sham tVNS); U value = 98.000

2. Secondary Outcome: Median Change From Baseline in Upper Extremity Fugl Meyer Assessment Score
Description: The median change in Upper Extremity Fugl-Meyer Score will be calculated from baseline to discharge at 3 weeks (immediately following the intervention) and again at 16 weeks (3 months follow-up from the intervention) in each training condition (sham tVNS + robotic arm training vs. active tVNS + robotic arm training). The median change in Upper Extremity Fugl Meyer score is reported, with a range 0-66 points, and with higher values indicating better functional status.
Time Frame: as for outcome 1
Population: 30 patients completed 9 sessions (3x/week for 3 weeks) of robotic arm training + sham or active tVNS, and 3 month follow-up at 16 weeks. A total of 30 participants were consequently included in the efficacy analysis.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Active tVNS + Robotic Arm Therapy | Sham tVNS + Robotic Arm Therapy
Number analyzed (Participants) | 15 | 15
scores on a scale
  Median change from baseline to discharge at 3 weeks | 2.000 [1.500 to 5.500] | 2.500 [1.500 to 4.500]
  Median change from baseline to 3 month follow-up | 2.330 [.0500 to 5.500] | 1.670 [1.000 to 4.500]
Statistical Analysis 1: Comparison: Active tVNS + Robotic Arm Therapy vs Sham tVNS + Robotic Arm Therapy; Test type: Equivalence — Statistical analysis of median change from baseline to DC immediately following 3 weeks of training was assessed with the upper extremity fugl meyer score in the active vs. sham tDCS conditions. Null hypothesis is that there is no difference in median change in upper extremity fugl meyer score between the active and sham tDCS conditions. A significance level of 0.05 was used (two-tailed); p = 1.000, Wilcoxon (Mann-Whitney) — The Mann-Whitney Wilcoxon test was performed to compare median change in Upper Extremity Fugl Meyer score from baseline to 3 weeks (discharge) across two separate study conditions (active vs. sham tVNS); U value = 112.000
Statistical Analysis 2: Comparison: Active tVNS + Robotic Arm Therapy vs Sham tVNS + Robotic Arm Therapy; Test type: Equivalence — Statistical analysis of median change from baseline to week 16 (3 month follow-up) was assessed with the Upper Extremity Fugl Meyer score in the active vs. sham tVNS conditions. Null hypothesis is that there is no difference in median change in Upper Extremity Fugl Meyer score between the active and sham tVNS conditions. A significance level of 0.05 was used (two-tailed); p = 0.950, Wilcoxon (Mann-Whitney) — The Mann-Whitney Wilcoxon test was performed to compare median change in Upper Extremity Fugl Meyer score from baseline to 16 weeks (follow-up) across two separate study conditions (active vs. sham tVNS); U value = 110.500

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for approximately 4 months, including the 3 week duration of the study intervention and the subsequent 3 month follow-up period.
Arm/Group | Active tVNS + Robotic Arm Therapy | Sham tVNS + Robotic Arm Therapy
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 2/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active tVNS + Robotic Arm Therapy (N=18) | Sham tVNS + Robotic Arm Therapy (N=18)
flu (Infections and infestations) | 0 (0) | 1 (1) — Subject suffered from the flu (unrelated to study intervention) and consequently missed repeated sessions. Subject was ultimately withdrawn from the study as a consequence.
wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Subject fractured wrist and was consequently unable to return for follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT03592745/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT03592745/ICF_001.pdf